CLINICAL TRIAL: NCT07248605
Title: Effect of Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices
Brief Title: Emergency Obstetric Care Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Nabil Ibrahim Mohamed, Nursing Specialist at specialized medical hospital -mansouraa uneversity hospital, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Applying Emergency Obstetric C
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Emergency Care; Obstetric

STUDY DESIGN:
Intervention Model Description: * The researcher will attend labor and delivery unit, emergency obstetric operating room and obstetric departments (9-10-15-18) at Mansoura University Hospital 3 days per week in cold days (Saturday, Monday and Wednesday) from 9:00 a.m. to 2:00 p.m. until the study sample is complete
  * The emergency obstetric care protocol will be carried out at pre-mentioned setting based on the results obtained from pre training assessment using the interviewing questionnaire and observational checklist.
  * Implementation of teaching and training will take (12) weeks. Nurses will be divided into (12) groups. Each group will include five nurses according to working circumstances and nurse's physical and mental readiness.
  * The overall sessions will be six sessions for each group divided into three theoretical sessions with a duration will be ranged from 30-45minutes for each, and three practical sessions while the duration of each practical session will be ranged from 30-60 minutes, The content will
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maternity nurses (Experimental): maternity nurses who are works in predetermined setting will be recruited except nurses who are on long vocations at the time of data collection or have administrative work.
  Interventions: Procedure: educational booklet

INTERVENTIONS:
Procedure: educational booklet — Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices

SUMMARY:
This study aims to investigate the effect of applying emergency obstetric care protocol on maternity nurses' practices.

DETAILED DESCRIPTION:
Effect of Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices Obstetrical emergencies are life threatening medical condition that occurs during pregnancy, labor or the postpartum period. Emergency Obstetric Care (EmOC) is categorized as Basic Emergency Obstetric Care (BEmOC) and Comprehensive Emergency Obstetric Care [CEmOC].

Treatments within BEmOC include the administration of parenteral antibiotics, oxytocics and anticonvulsants, manual removal of the placenta, removal of retained products of conception and assisted vaginal delivery. Comprehensive Emergency Obstetric Care (CEmOC) includes all of these plus blood transfusion and cesarean section.

The World Health Organization (WHO), 2020, posits the following conditions as obstetrical emergencies, ectopic or tubal pregnancy, abruptio placenta, placenta previa, sever preeclampsia & eclampsia or pregnancy induced hypertension, premature rupture of membranes, amniotic fluid embolism, inversion or rupture of uterus, placenta accreta, prolapsed umbilical cord, shoulder dystocia, postpartum hemorrhage and postpartum infection.

Globally, every year an estimated 287,000 women die of complications during pregnancy or childbirth. There are a variety of obstetrical emergencies of pregnancy that can threaten the well-being of both mother and newborn baby (WHO, 2019). Worldwide, obstetrical emergencies are the leading causes of maternal mortality particularly in developing countries where lack of transport facilities, financial constraints due to poverty, illiteracy, ignorance, inadequate health infrastructure and meager blood bank facilities.

Lack of nurse's knowledge and skills on how to recognize and manage obstetrical emergencies contribute to substandard institutional care and preventable maternal deaths (Kenya National Bureau of Statistics [KNBS] and International Coach Federation [ICF], 2023). Many studies have shown that health workers lack for the knowledge and skills to provide good quality care.

Proper knowledge about identification signs, emergency measures to be taken and a well-equipped obstetrics unit can reduce maternal mortality by almost 35- 40%, Maternity nurses are the main frontline skilled health personnel providing maternity care services globally. When educated, trained and regulated to national and international standards, maternity nurses can provide 90% of the needed essential care for women and newborns.

Most maternal complications are difficult to predict and prevent since any pregnant woman can develop them at any time during pregnancy, delivery or in the postpartum period (WHO, 2019). Thus, provision of effective, affordable and quality emergency obstetric care (EmOC) and efficient referral system plays pivotal role in promoting safe motherhood.

Immediate nursing management of the emergency cases is depending on the prompt action of the nurse and midwife recognition of the problem. She needs to recognize the onset of complications, perform intervention and practical skills that enables her to give emergency obstetrical care including life saving measures when needed being technically up-to-date on the latest evidence based skills and identifying those who are at the potential risk and referring them for expert care.

Although, pregnancy and childbirth is a normal process, complications may occur any time during antenatal or post natal period. Every delivery must be managed as an obstetrical emergency and all the preparation done to deal these emergencies. Skilled health professionals working in favorable environment should be available and able to attend to every pregnancy, delivery and must be available 24 hours a day, seven days a week.

Obstetrics emergency protocols are strategies geared towards reducing maternal deaths. The core elements of obstetrics emergency protocols include availability of skilled personnel to carry out effective interventions during pregnancy, delivery and postnatal period, availability of essential drugs and supplies and patient referrals.

The goals of emergency obstetric care protocol of critically ill women involve intensive monitoring and physiologic support for women with life-threatening to detect abnormal findings or subtle signs and symptoms of developing complications. Thus, the nursing contribution is very important to the rescue and mobilization of the team process to provide proper immediate care for the mother and the newborn and prevent any complication to be arises.

ELIGIBILITY:
Inclusion Criteria:

* of maternity nurses who are works in Obstetric departments , Emergency obstetric operating room and delivery unit

Exclusion Criteria:

* nurses who are on long vocations at the time of data collection or have administrative work.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices | after3 months of intervention
  Effect of Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices
Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices | after 3months of intervention
  Effect of Applying Emergency Obstetric Care Protocol on Maternity Nurses' Practices

CONTACTS AND LOCATIONS:
Overall Officials: Eman Nabil Ibrahim, doctor, Principal Investigator — Mansoura Uneversity; Eman Nabil Ibrahim, Principal Investigator — Specialist Nurse
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okonofua F, Ntoimo LFC, Ogu R, Galadanci H, Gana M, Adetoye D, Abe E, Okike O, Agholor K, Abdus-Salam RA, Randawa A, Abdullahi H, Daneji SM, Omo-Omorodion BI. Assessing the knowledge and skills on emergency obstetric care among health providers: Implications for health systems strengthening in Nigeria. PLoS One. 2019 Apr 8;14(4):e0213719. doi: 10.1371/journal.pone.0213719. eCollection 2019. PMID 30958834
- [Result] Brogaard L, Glerup Lauridsen K, Lofgren B, Krogh K, Paltved C, Boie S, Hvidman L. The effects of obstetric emergency team training on patient outcome: A systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2022 Jan;101(1):25-36. doi: 10.1111/aogs.14263. Epub 2021 Oct 8. PMID 34622945
- [Result] Amosse F, Boene H, Kinshella MW, Drebit S, Sharma S, Makanga PT, Vala A, Magee LA, von Dadelszen P, Vidler M, Sevene E, Munguambe K; Community Level Interventions for Pre-eclampsia (CLIP) Working Group. Implementation of a Community Transport Strategy to Reduce Delays in Seeking Obstetric Care in Rural Mozambique. Glob Health Sci Pract. 2021 Mar 15;9(Suppl 1):S122-S136. doi: 10.9745/GHSP-D-20-00511. Print 2021 Mar 15. PMID 33727325